CLINICAL TRIAL: NCT05073172
Title: A Randomized Intra-Patient Controlled Study of StrataXRT ® Versus Current Practice to Prevent and Treat Radiation Dermatitis
Brief Title: StrataXRT for the Prevention and Treatment of Radiation Dermatitis in Breast Cancer or Head and Neck Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study staff transition
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Josh Walker, M.D., Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00018789; NCI-2021-09431 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018789 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-09-16; First posted 2021-10-11 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Breast Carcinoma; Head and Neck Carcinoma; Radiation-Induced Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis | interventions — Petrolatum; Hydrogel, Polyethylene Glycol Dimethacrylate; Silver Sulfadiazine; Hydrocortisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (StrataXRT) (Experimental): Patients apply StrataXRT topically to the affected area once or twice daily starting from the first dose of radiation therapy until dermatitis has returned to grade =< 1.
  Interventions: Drug: Silicone-based Film Forming Topical Gel
- Arm II (standard of care) (Active Comparator): Patients receive standard of care including calendula and/or Aquaphor applied 2-6 times daily plus hydrogel or Silvadene or topical corticosteroids applied twice daily starting from the first dose of radiation therapy until dermatitis has returned to grade =< 1.
  Interventions: Drug: Calendula Ointment; Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment; Other: Polyethylene Glycol Hydrogel; Drug: Silver Sulfadiazine; Drug: Topical Hydrocortisone

INTERVENTIONS:
Drug: Calendula Ointment — Applied topically
  Arms: Arm II (standard of care)
Other: Petrolatum-Mineral Oil-Lanolin-Ceresin Ointment — Applied topically
  Other Names: Aquaphor
  Arms: Arm II (standard of care)
Other: Polyethylene Glycol Hydrogel — Applied topically
  Other Names: PEG Hydrogel
  Arms: Arm II (standard of care)
Drug: Silicone-based Film Forming Topical Gel — Applied topically
  Other Names: Silicone-based Film-forming Gel Dressing; StrataCTX; StrataXRT; StrataXRT Gel
  Arms: Arm I (StrataXRT)
Drug: Silver Sulfadiazine — Applied topically
  Other Names: Flamazine; Silvadene; Sliverex; SSD; Sulfadiazine Silver; Thermazene
  Arms: Arm II (standard of care)
Drug: Topical Hydrocortisone — Applied topically
  Arms: Arm II (standard of care)

SUMMARY:
This clinical trial studies the effect of StrataXRT in preventing and treating radiation dermatitis in breast cancer or head and neck cancer patients. Radiotherapy is often associated with multiple side effects. These side effects can cause patient injury and make it difficult to complete treatment. For example, radiation dermatitis or skin damage may result in severe skin peeling and skin irritation. Depending on the location of radiation, the skin damage can cause problems and be tough to heal. This trial aims to see whether StrataXRT may help to prevent dermatitis after radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare efficacy of silicone-based film forming topical gel (StrataXRT) versus (vs.) standard of care skin maintenance.

SECONDARY OBJECTIVES:

I. Evaluate overall effectiveness of StrataXRT. II. Evaluate post-radiation therapy (RT) recovery time for StrataXRT compared to standard of care.

EXPLORATORY OBJECTIVES:

I. To assess patient reported outcomes. II. Evaluate cost of StrataXRT for management of radiation dermatitis compared to standard of care skin maintenance.

III. Evaluate the reduction in RT interruption/extension of overall duration of receiving RT based on the reduced skin toxicity.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients apply StrataXRT topically to the affected area once or twice daily starting from the first dose of radiation therapy until dermatitis has returned to grade =< 1.

ARM II: Patients receive standard of care including calendula and/or petrolatum-mineral oil-lanolin-ceresin ointment (Aquaphor) applied 2-6 times daily plus hydrogel or silver sulfadiazine (Silvadene) or topical corticosteroids applied twice daily starting from the first dose of radiation therapy until dermatitis has returned to grade =< 1.

After completion of study, patients are followed up at 6 days and 3 weeks post-RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be adult (> age of 18) patients. Both men and women and members of all races and ethnic groups will be included
* Histologically confirmed malignancy for which standard curative measures in conjunction with radiotherapy are indicated to the following sites: whole breast/chest-wall for post-surgical radiotherapy or bilateral neck (levels one through six) for head and neck cancer
* All head and neck cancer patients should have the left and right neck treated to the same dose when receiving bilateral neck irradiation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Clinically evident skin involvement of malignancy
* Thin patients with nodal involvement requiring bolus
* Patients with significant unshaven facial or chest wall hair compromising film application
* Evidence of active cellulitis or wound infection involving anticipated treatment site
* History of prior radiotherapy to involved site within 5 cm of anticipated treatment field
* Eastern Cooperative Oncology Group (ECOG) performance status >= 3
* Patients receiving concurrent capecitabine
* Patient with skin grafts over treatment site(s)
* Presence of psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. (i.e. schizophrenia, autism, temporary housing during treatment, scheduling conflict immediately after treatment. This will need to be assessed prior to consent
* Actual or perceived inability to reliably apply StrataXRT to the patients treatment field in the home environment
* Anticipated or actual use of other non-study topical medications or remedies in the treatment field
* Vulnerable populations (pregnant women, decisionally impaired adults, and prisoners) will be excluded from the study
* Patients receiving ultra-hypofractionated radiation to the breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Radiation dermatitis | Day 0 post-radiation therapy (RT)
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Grade 2+ radiation dermatitis | Day 0 post-RT
  Will be assessed by CTCAE version 5.0.
Grade 2+ radiation dermatitis | Day 6 +/- 1 post-RT
  Will be assessed by CTCAE version 5.0.
Weekly Common Terminology Criteria for Adverse Events (CTCAE) scores | Up to week 3 post-RT
  Will continue to assess CTCAE score for radiation dermatitis until resolution of symptoms.
Time to peak Common Terminology Criteria for Adverse Events (CTCAE) score | Up to week 3 post-RT
Post-RT recovery time (to grade =< 1 radiation dermatitis | Up until entire irradiated treatment site healed (grade =< 1 dermatitis)
  Will be defined by Common Terminology Criteria for Adverse Events (CTCAE).

OTHER OUTCOMES:
Weekly Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) scores | Up to week 3 post-RT
Average cost of StrataXRT tubes | Until healed (grade =< 1 dermatitis), up to 10 weeks
Incidence of use of skin care products in addition to StrataXRT | Until healed (grade =< 1 dermatitis), up to 10 weeks
Overall RT duration | Up to Day 0 post-RT
Number of days missed (attributable to patient or provider concern re: dermatologic toxicity) | Up to Day 0 post-RT

CONTACTS AND LOCATIONS:
Overall Officials: Josh Walker, M.D., Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States